CLINICAL TRIAL: NCT03514849
Title: Clinical Study of Combined Radical Operation With Postoperative Adjuvant Chemotherapy and Prophylactic Cranial Irradiation in pT1-2N0M0 Stage of Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peng Zhang (Other)
Responsible Party: Sponsor-Investigator, Peng Zhang, Director of science and education, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k18-065
Record Dates: First submitted 2018-04-11; First posted 2018-05-02 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI group (Experimental)
  Interventions: Procedure: prophylactic cranial irradiation (PCI); Procedure: lobectomy + mediastinal lymph node dissection or systematic lymph node sampling; Drug: postoperative adjuvant chemotherapy
- Control group (Placebo Comparator)
  Interventions: Procedure: lobectomy + mediastinal lymph node dissection or systematic lymph node sampling; Drug: postoperative adjuvant chemotherapy

INTERVENTIONS:
Procedure: prophylactic cranial irradiation (PCI) — Patients in the control group are enrolled in the follow-up, and the patients in research group will receive prophylactic cranial irradiation （PCI） by 25 gy/10 fx.
  Arms: PCI group
Procedure: lobectomy + mediastinal lymph node dissection or systematic lymph node sampling — lobectomy + mediastinal lymph node dissection or systematic lymph node sampling
Drug: postoperative adjuvant chemotherapy — If the postoperatively pathological examination of the patient is confirmed to be in pT1-2N0 stage, a single postoperative adjuvant chemotherapy (combining etoposide with cisplatin) is recommended. If patients are difficult to tolerate the side effects of cisplatin, we can replace cisplatin by carboplatin in the adjuvant chemotherapy scheme.

SUMMARY:
At present, for participants with cT1-2N0 small cell lung cancer (SCLC), the International guidelines recommend surgical radical resection (lobectomy + systematic lymph node sampling or cleaning); If the postoperatively pathological examination is confirmed to be in pT1-2N0 stage, a single postoperative adjuvant chemotherapy (combining etoposide with cisplatin) is recommended. If participants are difficult to tolerate the side effects of cisplatin, the investigators can replace cisplatin by carboplatin in the adjuvant chemotherapy scheme. Participants with pT1-2N0 SCLC are not recommended to receive postoperative chest-assisted radiotherapy. For participants with pT1-N0 SCLC after specific surgical resection, prophylactic cranial irradiation (PCI) is currently recommended. But this recommendation is currently lacking the support of research evidence.

The main purpose of this study is to study the prognostic effects of PCI on participants with pT1-2N0 stage small cell lung cancer (SCLC) who have received radical surgery and postoperative adjuvant chemotherapy.

The main endpoint of this study is to observe the total survival rate (5-year OS%) in 5 years.

The secondary outcome measures include 5 years of disease-free survival (5-year DFS%), disease-free survival (DFS), overall survival (OS), surgical complications, resection rates, quality of life (QoL), and exploration of biomarkers (tumor tissue).

This is a two-arm, open, multicentral clinical study designed to compare the 5-year OS% of participants receiving or not receiving PCI for pT1-2N0 stage small cell lung cancer (SCLC) with radical surgery plus postoperative adjuvant chemotherapy. Previous literature reports that the 5-year OS% of participants with pT1-2N0 period SCLC who have received surgical resection is about 50%. Assuming that PCI can increase 5 years OS% by 10%, then enrolling 320 participants in the group can guarantee 70% degree of certainty with observing a unilateral significant difference α< 0.1. Taking about 10% of the follow-up loss rate into account, the investigators expect to enroll 360 participants.

Dividing the 360 participants divided into two groups randomly, each group is composed of 180 people. All participants received lobectomy plus mediastinal lymph node dissection or systematic lymph node sampling. Participants in the control group are enrolled in the follow-up, and the participants in research group will receive PCI by 25gy/10fx.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Ability to follow research programs and follow-up procedures;
* * Patient age ≥ 18 years old;
* Histology or cytology confirmed as SCLC, chest enhancement ct, liver and adrenal ct, skull MRI, pet-ct/whole body bone scintigraphy, ebus puncture biopsy, etc. clearly as the t1-2n0 period of the initial treatment of patients (according to the UICC 2009 version of the phased standard);
* Radical resection of the leaf, the postoperative confirmed margin negative, pathological stage of t1-2n0 stage of small cell lung cancer;
* 4-week EP or EC regimen for adjuvant chemotherapy after surgery;
* Physical status ECOG assessment is divided into 0~1;
* Life expectancy at least 12 weeks;
* The following laboratory tests conducted within 21 days of the end of the 4th cycle of chemotherapy confirmed that the patient's bone marrow, liver and kidney function met the requirements for participation in the study:
* Hemoglobin ≥9.0 g/dl (can be maintained or exceeded by blood transfusion);-Neutrophil absolute Count (ANC) ≥1.5x109;
* Platelet count ≥100x109/mm3;
* Total bilirubin ≤ 1.5 times times normal value upper limit;
* Alt and Straw transaminase ≤ 2.5 times times the normal value of the upper limit;
* creatinine ≤ 1.5 times times the upper limit of normal value and creatinine clearance rate ≥60ml/min; -prothrombin Time International standardized ratio (INR) ≤1.5, and part of the clotting activity Time (APTT) ≤ 1.5 times times the normal value limit.
* Patients who received a full or parenteral anticoagulation treatment had a minimum dose of anticoagulant for at least 2 weeks before entering clinical studies, and the results of the coagulation test were available for clinical trials within the limits of local treatment.
* Women of childbearing age must be tested in pregnancy for 7 days prior to initiation of treatment and negative results.
* Men and women of the appropriate age are required to use a reliable method of contraception until 30 days after withdrawal from the study before entering the trial. Reliable contraceptive methods will be judged by the principal researcher or designated person.

Exclusion Criteria:

* Patients who have conducted any systemic anticancer therapy for SCLC, including cytotoxic drug therapy, targeted drug therapy and experimental therapy.
* Localized radiotherapy for SCLC;
* Patients with cancer other than SCLC in the five years prior to the start of the study.
* Except for cervical in situ carcinoma, cured basal cell carcinoma, bladder epithelial tumor [including TA and tis];
* Any unstable systemic disease (including active infections, uncontrolled high blood pressure, unstable angina pectoris, onset of angina in the last 3 months, congestive heart failure (≥ "NYHA" Grade II), cerebral infarction (6 months before the group), severe arrhythmia requiring medical treatment, Diagnosis with liver, kidney or metabolic disease;
* Has or is currently suffering from interstitial lung disease;
* Lack of full control of ocular inflammation or eye infections, or any condition that may cause such ocular diseases;
* Known human immunodeficiency virus (HIV) infection;
* Allergy to any kind of research drug;
* Patients undergoing major surgery or severe trauma within 2 months prior to the first medication;
* any negative absorption;
* Pregnant or lactating women;
* Other researchers do not think fit into the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival rate(5-y OS%) | From the completion of the intervention to 5 years.
  Five-year survival rate measures survival at 5 years after surgery.

SECONDARY OUTCOMES:
5-year disease-free survival rate (5-y DFS%) | From the completion of the intervention to 5 years.
  The rate that the patients whose disease doesn't recur take up in the total patients from the start of randomization to 5 years.
disease-free survival period | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  From the beginning of randomization to the time-point when the disease recurs or the patient dies due to disease progression.
overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Patients die directly from the progression of SCLC or from an unrelated cause (for example, a car accident). When the precise cause of death is not specified, this is called the overall survival rate.
surgery complications | Within 2 weeks includes surgery and perioperative period.
  The complications related to the operations that happen in the perioperative period.
removal rate | Through study completion, an average of 1 year.
  The patients who are able to receive the radical resection.
tumor biological makers | Within 2 weeks includes surgery and perioperative period.
  To search the possible bio-makers for SCLC.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided